CLINICAL TRIAL: NCT05728060
Title: Associations of Fecal Bile Acid Profile and Intestinal Flora With Chronic Radiation Enteritis
Status: Completed | Type: Observational
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Principal Investigator, Clinical Professor, Xijing Hospital of Digestive Diseases
Other Study IDs: KY20222208-F-1
Record Dates: First submitted 2023-02-04; First posted 2023-02-14 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Radiation Enteritis
Keywords: Radiation Enteritis; Bile Acid; Gut Microbiota

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Fecal samples will be stored in liquid nitrogen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- chronic radiation enteritis: Non-surgically treated cervical cancer patients develop chronic radiation enteritis after radiation therapy.
- No chronic radiation enteritis after radiotherapy: Patients with non-surgical cervical cancer do not develop chronic radiation enteritis after radiation therapy.
- Patients with cervical cancer: Patients with cervical cancer did not undergo any treatment.

SUMMARY:
To explore the fecal bile acid profile of patients with radiation enteritis, to clarify the types of bile acids that are closely related to the occurrence of radiation enteritis; to explore the interaction between fecal bile acids and intestinal flora in patients with radiation enteritis, and to lay the foundation for further elucidation of the pathogenesis of radiation enteritis.

ELIGIBILITY:
Inclusion Criteria:

1. . non-surgical cervical cancer patients aged 18 to 75 years who received radiotherapy;
2. . Patients who can fully understand the content of informed consent for this trial and voluntarily sign the written informed consent;
3. . able to receive follow-up examinations, follow-up examinations, and specimen retention on time;
4. . The case group met the diagnostic criteria for chronic radiation enteritis in the "Expert Consensus on the Diagnosis and Treatment of Radiation Proctitis in China (2018 edition)"; Control group 1: Non-surgical cervical cancer patients without chronic radiation enteritis after radiotherapy; Control group 2: Patients with cervical cancer who did not receive any treatment.

Exclusion Criteria;

1. . Presence of diseases affecting bile acid metabolism, such as hepatitis and cirrhosis of the liver from various causes, gallstones, etc;
2. . Patients who have previously undergone cholecystectomy or partial resection of the intestine;
3. . Taking drugs affecting bile acid metabolism due to other diseases, such as cholestyramine, anti-inflammatory and Xiaoyan lidan tablets, Danshu capsules, ursodeoxycholic acid, obeticholic acid, and proprietary Chinese medicines such as schisandrin B, Tanshinone IIA, and Yinjiazhuang;
4. . Recent use of drugs that affect gastrointestinal motility;
5. . Patients with moderate or severe renal impairment (blood creatinine > 2 mg/dL or 177 mmol/L), or abnormal liver function (ALT > 2 times the upper limit of normal value); moderate or severe chronic obstructive pulmonary disease; patients with severe hypertension, patients with cerebrovascular accidents; patients with congestive heart failure, unstable angina pectoris;
6. . Patients with mental or legal disabilities;
7. . Suspected or confirmed history of alcohol/substance abuse or other pathology that, in the judgment of the investigator, reduces the likelihood of enrollment or complicates enrollment;
8. . Refuse to sign informed consent;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients are from Xijing Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Correlation between fecal bile acid profile and chronic radiation enteritis | 7 months
  Patients' fecal bile acid profiles were analyzed by ultra-performance liquid chromatography-tandem mass spectrometry and screened for the bile acids associated with chronic radiation enteritis.

SECONDARY OUTCOMES:
Correlation between fecal bile acid profile and intestinal microbiota in different groups. | 7 months
  Investigators explore the cross-talk between fecal bile acid and gut microbiota according to the results of 16s rRNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, PhD, Study Director — Xijing Hosipital of Digestive Disease
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Shen X, Li SB, Gao MJ, Cao JJ, Yang H, Li WW, Wei LC, Chen M, Liu JY, Shi YQ. Relationship Between Fecal Bile Acid Profile and Intestinal Microbiota in Patients With Chronic Radiation Enteritis. J Dig Dis. 2026 Jan 28. doi: 10.1111/1751-2980.70029. Online ahead of print. PMID 41605669